CLINICAL TRIAL: NCT05626192
Title: Anatomical Evaluation of the APL and FCR Tendons in Thumb CMC Joint in Relation to Osteophytes Formation of the Trapezium and Osteoarthritis.
Brief Title: Anatomical Evaluation of the APL Tendons in Thumb CMC Joint and Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CMC-2022-69
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-09

CONDITIONS: Thumb Osteoarthritis
Keywords: Thumb Osteoarthritis; Enthesis organ; Sensory nerve endings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Anatomical dissection and Immunohistochemical techniques — Anatomical dissection and description

SUMMARY:
Certain ligaments in the human body are designed to be a static stabilizer and others to have a sensory function thus remains an unresolved issue.

The presence of mechanoreceptors (sensory corpuscles and free nerve endins) in the human knee and ankle ligaments has implies a sensory role of ligaments in providing afferent information, which in turn regulates intrinsic stiffness in the muscles surrounding the joint, contribuiting to dynamic joint stability.

The aim of this study is to use immunohistochemical methods to analyze the general innervation and possible existence of sensory corpuscles in the thumb carpometacarpal (CMC) joint. This study can help to know the contribution of the tendon insertions and ligaments in the dynamic thumb CMC joint stability.

DETAILED DESCRIPTION:
The accessory APL tendons insertions, number of accessory tendons and insertion in trapezium can be a mechanical factor that develop osteophytes and thumb CMC joint osteoarthritis.

Antibodies against the general nerve marker protein gene product 9.5 (PGP 9.5) and the glial marker S-100 will be use to depict innervation and corpuscular structures. Innervation pattern and sensory corpuscules were investigated by other authors in the wrist. S-100 immunoreactivity is in the Schwann cells in the central regions of the corpuscle, and PGP 9.5 immunoreactivity marked the axonal structures in the corpuscles. The presence of nerve fascicles and particularly sensory corpuscles in the structures, for exemple capsule and APL insertion near the thumb carpometacarpal joint suggest that these structures in the CMC joint have a propioceptive role in the stability of the joint.

ELIGIBILITY:
Inclusion Criteria:

* Specimens: Adults from 50 to 90 years.

Exclusion Criteria:

* Specimens: younger than 50 or older than 90 years.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study will include 20 specimens. The first part of the study will be a dissection of the specimens. Description of the variability of tendons in the first extensor compartment. The investigators analyze the APL tendon insertion, osteophytes formation and osteoarthritis in thumb CMC joint . In the second part of the study, the researchers will take a small sample of the APL insertion with the osteophyte, capsule and ligaments in the thumb CMC joint. The investigators will fix the sample in a solution of 4% formaldehyde and they will stain the samples with hematoxylin eosin. Immunohistochemistry with PGP 9.5 and S-100.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-11-13 (Actual); Primary Completion 2024-08-16 (Estimated); Study Completion 2024-12-23 (Estimated)

PRIMARY OUTCOMES:
Number of APL tendon insertions in trapezium in thumb CMC joint | 12 months
  Description of the distribution of the APL tendons in thumb CMC joint. Measure in number from 1 to 10 insertions.
Osteophytes formation and thumb CMC joint osteoarthritis (OA) | 12 months
  Thumb carpometacarpal joint osteoarthitis and osteophytes. Classifying the thumb OA in the specimens according to the International Cartilage Repair Society (ICRS) cartilage lesion classification system. Measure of the loss of cartilage in the CMC joint surface in millimeters (mm) with a digital caliper.

SECONDARY OUTCOMES:
Sensory nerve endings and mechanoreceptors in thumb CMC joint | 12 months
  Analyze the types of sensory nerve endings and mechanoreceptors in thumb CMC joint using immunohistochemical techniques: hematoxylin eosin , S100, PGP-95, in order to gain more insight into functional CMC joint stability. Measure in number from 0 to 20 sensory nerve endings.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lamas, MD, Ph D, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Claudia Erika Delgado Espinoza, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: No
Protocol for the collection of anatomical variants of the APL tendon insertions and the association with osteophytes formation and thumb CMC joint osteoarthritis.

REFERENCES:
- [Result] Adams JE, O'Brien V, Magnusson E, Rosenstein B, Nuckley DJ. Radiographic Analysis of Simulated First Dorsal Interosseous and Opponens Pollicis Loading Upon Thumb CMC Joint Subluxation: A Cadaver Study. Hand (N Y). 2018 Jan;13(1):40-44. doi: 10.1177/1558944717691132. Epub 2017 Feb 16. PMID 28719976
- [Result] Choi SY, Rhim J, Han WJ, Park H, Noh JW, Han J, Ha CW. Associations between biomarkers and histological assessment in individual animals in a destabilization of the medial meniscus (DMM) model of osteoarthritis (OA). Acta Orthop Belg. 2021 Dec;87(4):713-721. doi: 10.52628/87.4.16. PMID 35172438
- [Result] Deivasigamani S, Azad A, Yang SS. The Variable Insertional Anatomy of the Abductor Pollicis Longus: Functional Relevance and Relationship to Adjacent Thumb Extensors. Hand (N Y). 2023 Jan;18(1):145-152. doi: 10.1177/1558944721999734. Epub 2021 Apr 1. PMID 33789520
- [Result] Gupta S, Michelsen-Jost H. Anatomy and function of the thenar muscles. Hand Clin. 2012 Feb;28(1):1-7. doi: 10.1016/j.hcl.2011.09.006. PMID 22117918
- [Result] Freeman MA, Wyke B. The innervation of the ankle joint. An anatomical and histological study in the cat. Acta Anat (Basel). 1967;68(3):321-33. doi: 10.1159/000143037. No abstract available. PMID 5591904
- [Result] Hagert E, Lee J, Ladd AL. Innervation patterns of thumb trapeziometacarpal joint ligaments. J Hand Surg Am. 2012 Apr;37(4):706-714.e1. doi: 10.1016/j.jhsa.2011.12.038. PMID 22464234
- [Result] Hagert E, Garcia-Elias M, Forsgren S, Ljung BO. Immunohistochemical analysis of wrist ligament innervation in relation to their structural composition. J Hand Surg Am. 2007 Jan;32(1):30-6. doi: 10.1016/j.jhsa.2006.10.005. PMID 17218173
- [Result] Hagert E, Ljung BO, Forsgren S. General innervation pattern and sensory corpuscles in the scapholunate interosseous ligament. Cells Tissues Organs. 2004;177(1):47-54. doi: 10.1159/000078427. PMID 15237195
- [Result] Kofman KE, Schuurman AH, Mulder MC, Verlinde SA, Gierman LM, van Diest PJ, Bleys RL. The pisotriquetral joint: osteoarthritis and enthesopathy. J Hand Microsurg. 2014 Jun;6(1):18-25. doi: 10.1007/s12593-014-0129-3. Epub 2014 Apr 18. PMID 24876685
- [Result] Ladd AL, Lee J, Hagert E. Macroscopic and microscopic analysis of the thumb carpometacarpal ligaments: a cadaveric study of ligament anatomy and histology. J Bone Joint Surg Am. 2012 Aug 15;94(16):1468-77. doi: 10.2106/JBJS.K.00329. PMID 22992815
- [Result] McGee C, O'Brien V, Van Nortwick S, Adams J, Van Heest A. First dorsal interosseous muscle contraction results in radiographic reduction of healthy thumb carpometacarpal joint. J Hand Ther. 2015 Oct-Dec;28(4):375-80; quiz 381. doi: 10.1016/j.jht.2015.06.002. Epub 2015 Jun 27. PMID 26209165
- [Result] Menz HB, Marshall M, Thomas MJ, Rathod-Mistry T, Peat GM, Roddy E. Associations Between Calcaneal Enthesophytes and Osteoarthritis of the Hands and Feet. Arthritis Care Res (Hoboken). 2020 Oct;72(10):1343-1348. doi: 10.1002/acr.24030. PMID 31325208
- [Result] Moriggl B, Kumai T, Milz S, Benjamin M. The structure and histopathology of the "enthesis organ" at the navicular insertion of the tendon of tibialis posterior. J Rheumatol. 2003 Mar;30(3):508-17. PMID 12610810
- [Result] Opreanu RC, Wechter J, Tabbaa H, Kepros JP, Baulch M, Xie Y, Lackey W, Katranji A. Anatomic variations of the first extensor compartment and abductor pollicis longus tendon in trapeziometacarpal arthritis. Hand (N Y). 2010 Jun;5(2):184-9. doi: 10.1007/s11552-009-9234-3. Epub 2009 Oct 16. PMID 19834771
- [Result] Rein S, Hagert E, Hanisch U, Lwowski S, Fieguth A, Zwipp H. Immunohistochemical analysis of sensory nerve endings in ankle ligaments: a cadaver study. Cells Tissues Organs. 2013;197(1):64-76. doi: 10.1159/000339877. Epub 2012 Sep 4. PMID 22964904
- [Result] Rein S, Krenn V, Hagert E, Garcia-Elias M, Lluch A, Kremer T, Semisch M. Degeneration of the articular disc in the human triangular fibrocartilage complex. Arch Orthop Trauma Surg. 2021 Apr;141(4):699-708. doi: 10.1007/s00402-021-03795-2. Epub 2021 Feb 6. PMID 33550482
- [Result] Wu Z, Nagata K, Iijima T. Involvement of sensory nerves and immune cells in osteophyte formation in the ankle joint of adjuvant arthritic rats. Histochem Cell Biol. 2002 Sep;118(3):213-20. doi: 10.1007/s00418-002-0443-x. Epub 2002 Jul 19. PMID 12271357